CLINICAL TRIAL: NCT04932408
Title: Evaluation of the Feasibility, Psychosocial Effects, Influence and Perception of Exercise Selection and Experimental Design of Exercises Performed.
Brief Title: The Feasibility of a Dynamic Exercise Intervention. Psychosocial Effects and Process Evaluation of the Experimental Design.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Derby (Other)
Responsible Party: Principal Investigator, Nichola Davis, Principal Investigator: Miss Nichola Michelle Davis (PhD Student), University of Derby
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UDerby
Record Dates: First submitted 2021-06-06; First posted 2021-06-21 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Stability; Old Age; Debility; Balance; Distorted
MeSH Terms: conditions — Frailty | interventions — Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hip Region (Experimental): Pre selected exercises (8) will be performed by the participant using an elastic resistance band anchored from ground level and placed around the hip region.
  Warm up: 5-10 mins
  Exercises:
  Forward step, forward tandem steps, forward tandem hold, Upper body rotation, side steps. backward step, backward tandem walk, backward tandem hold.
  Cool down. Post intervention- Semi-structured Interview schedule
  Interventions: Other: Evaluation of the feasibility, psychosocial effects, influence and perception of exercise selection an experimental design of exercises performed at the hip and chest region.
- Chest Region (Experimental): Pre selected exercises (8) will be performed by the participant using an elastic resistance band anchored from ground level and placed the chest region (using velcro on a chest harness/training vest).
  Warm up: 5-10 mins
  Exercises:
  Forward step, forward tandem steps, forward tandem hold, Upper body rotation, side steps. backward step, backward tandem walk, backward tandem hold.
  Cool down. Post intervention- Semi-structured Interview schedule
  Interventions: Other: Evaluation of the feasibility, psychosocial effects, influence and perception of exercise selection an experimental design of exercises performed at the hip and chest region.

INTERVENTIONS:
Other: Evaluation of the feasibility, psychosocial effects, influence and perception of exercise selection an experimental design of exercises performed at the hip and chest region. — A single exposure feasibility study using elastic resistance bands in older adults to challenge stability. Exercises with an elastic resistance band anchored from the ground and placed at the hip and chest region will be trialled. A semi- structured interview will identify the impact and practicalities of the intervention. The information will be used in the development of an evaluation process with key consideration of the planning phase of the intervention. Questions with verbal cues to provide perceptions of the exercise selection such as likes/dislikes, safety, confidence, difficulty, enjoyment and band placement will be asked to determine the acceptability, accessibility, appropriateness and usability of the protocol and build insights into the participant preferences.
  Other Names: Elastic Resistance Band Training; Balance training in Older Adults; Stability Training using Resistance bands in Older Adults; The feasibility of using Elastic Resistance Bands in Older Adults; Novel Elastic Resistance Band training Intervention in Older Adults; Feasibility study on a Novel Elastic Resistance Band training Intervention

SUMMARY:
Current balance and stability interventions have been shown to improve balance through targeting balance impairments and retraining effects. However, there are key facilitators and barriers 'that older adults may face to participate in such interventions'. Additionally, physical activity interventions fail to integrate older adults into the co-design and co-production of PA interventions.

The study will aim to identify the impact and practicalities of an exercise intervention in older adults by performing pre selected exercises with an elastic resistance band attached at the hip and chest region to challenge balance. Researcher led interviews will focus on the participants perceptions of the activities and decision making of exercise selection by selecting components that they are confident to perform which is a key element to creating a practical and enjoyable exercise programme for the older population. This will co-create an intervention that is accessible, acceptable, and appropriate for older adults.

The study will establish the accessibility, acceptability and appropriateness of an elastic band exercise intervention with older adults by performing selected activities followed by researcher led interviews that will focus on the participants influences, perceptions and psycho-social factors related the intervention activities.

DETAILED DESCRIPTION:
Outline of study design The following study will be designed as a single exposure, qualitative (one-to-one interviews using a semi-structured interview guide) and quantitative (heart rate and rate of perceived exertion ratings) study. A convenience sample of adults/older adults will be recruited through PA networks in the Derbyshire community. Participants will take part in one experimental session: performing exercises with an elastic resistance band placed at the hip and chest region. The session order of band placement will be randomized for each participant to counter-balance the outcome which emerge from the study.

Participant preparation Following a detailed briefing using a pre-prepared participant information sheet, a signed informed consent form and Instrumental Activities of Daily Living form, participants will be required to complete 2 supervised visits to the laboratory at the University of Derby.

Participants will complete a general health screening questionnaire. Specific instructions will be provided for participants to abstain from alcohol and caffeine for a minimum of 12/24 hours respectively and avoidance of strenuous exercise for at least 72 hours prior to participation.

Outline of study methods Participants will be required to attend the University Laboratory (Kblock) to take part in the study. Due to COVID-19 participants will be required to adhere to the latest government guidance and guidance from the University to consider this assessment to be safe (Risk assessments in place).

Baseline assessments:

* Mini Balance Evaluation (MINI BESTest)
* Short Falls Efficacy Scale (Short FES-I)

Following a briefing, participants will be required to perform a 10 minute supervised warm up and mobility session prior to exercise. Participants will be required to perform a selection of 8 pre-selected exercises whilst wearing the elastic band around the hip or chest region (randomized) with a 20 minute rest in between each condition). Participants will perform the exercises with the lowest resistance of 2-15lb aimed at low/moderate intensity. Heart rate (HR) on a heart rate strap and watch, rate of perceived exertion (RPE) (Borg scale) will be measured to assess exercise intensity.

All sessions will be closely supervised by the lead researcher -a qualified postural stability instructor, (level 4 reps Postural Stability Instructor trained by Later Life Training), that will provide prompts on form of the exercises.

Elastic band placement

Hip region:

Each participant will be required to perform the series of exercises whilst attached to an elastic resistance band. The elastic band will be attached from ground level which will be attached to the participant over the hip region with padding.

Chest region Each participant will be required to perform a series of exercises whilst attached to an elastic resistance band. The elastic band will be attached from ground level and to the participant over the chest region (under arms) , using Velcro on a chest harness/training vest.

Immediately following the single-session exercise intervention, participants will be required to attend a one-on-one, face to face semi-structured interview with the researcher to identify the impact and practicalities of the exercise intervention. The information will be used in the development of an evaluation process with key consideration of the planning phase of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be male and females over 50 years old. Although ageing is an individual and qualitative perspective rather than solely a chronological perspective, adults are transitioning to older adulthood in their 5th decade of life. Older adults may benefit from preparing at an earlier stage of ageing from the age of 50 years compared to beginning at the age of 65 years where falls are a high risk factor. PA guidelines recommend that adults will benefit from preparing physical attributes such as strength and balance at an earlier stage of the ageing process, therefore, this age group of 50 years and over has been selected as the most appropriate.
* Moderately Physically active (this will be determined by the International Physical Activity Questionnaire (IPAQ) prior to participation of the study. A score of at least 600 MET-min/week (moderate physical activity level) will be required to take part in the study.
* Ability to walk without a walking aid
* Ability to provide consent. This will be determined by using the Mini-Mental State Examination (MMSE) a score of under 23. The MMSE will assess cognitive function using scoring to ensure that participants are not cognitively impaired

Exclusion Criteria:

* Individuals that are under the age of 50 years old
* Individual that have serious, unstable cardiovascular conditions such as recent acute myocardial infarction; congestive heart failure; uncontrolled hypertension; serious musculoskeletal or neurologic conditions (including Parkinson's disease, Huntington's disease, acute stroke, paresis of the lower limbs and uncontrolled diabetes mellitus.
* Individuals with acute respiratory tract infection or chronic lung disease (e.g. asthma and obstructive pulmonary disease).
* Individuals that are not physically active (METs score under 600 MET-min/week). have severe cognitive impairment (inability to follow simple training instructions; and acute respiratory tract infection or chronic lung disease (e.g. asthma and obstructive pulmonary disease).
* Individuals that are unable to provide consent. This will be determined by using the Mini-Mental State Examination (MMSE)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Semi structured Interview | through study completion, an average of 1 year
  A one-on-one, face to face semi-structured interview with the researcher to identify the impact and practicalities of the exercise intervention. The information will be used in the development of an evaluation process with key consideration of the planning phase of the intervention. A semi-structured interview schedule developed by the lead researcher will investigate the acceptability, accessibility, appropriateness and usability of the protocol. Participants will be asked a series of open and closed questions and likert scales to provide perceptions of the exercise selection such as likes/dislikes, safety, confidence, difficulty, enjoyment and band placement. This will help to build insights into the participant preferences which is an important element of the intervention design.
Heart rate | through study completion, an average of 1 year
  Heart rate measures will be taken during each exercise. Higher values = higher exertion of each exercise performed. 50 beats per min - 120 = low, 120- 150 beats per min = moderate and 150 beats per min = high.
Rate of perceived exertion (RPE) | through study completion, an average of 1 year
  RPE measures will be taken during each exercise. Scale 0-10. 0= no exertion and 10 being the highest exertion- exhaustion.

SECONDARY OUTCOMES:
Mini Balance Evaluation Test (MINI-BESTest) | through study completeion, an average of 1 year
  This assessment will require participants to perform a series of physical performance tasks. Following each task, the researcher will record the scores to sum a total score for the MINI BESTest. Scoring: The test has a maximum score of 28 points from 14 items that are each scored from 0-2. "0" = lowest level of function and "2" = highest level of function.
  If a subject must use an assistive device for an item, score that item one category lower.
  If a subject requires physical assistance to perform an item, score "0" for that item.
Short Falls efficacy scale | through study completion, an average of 1 year
  This questionnaire will require the participant to answer 7 questions on their own perceptions on concerns of falling during a series of activities. The scale for each questions is measured from a value of 1-4. 1 = not concerned at all about falling and a 4 =very concerned about falling for each item. A higher score on the FES-l will represent a greater concern for falls from a participant (lowest score 7 and highest score 28).

OTHER OUTCOMES:
Instrumental Activities of Daily Living form (IADL) | through study completion, an average of 1 year
  To identify how a person is functioning at the present time to determine any differences in participation recruitment. The IADL has 8 categories which the participant is required to select one out of four options that have a score assigned to their level of functioning (either 1 or 0). Scoring Interpretation: In some activities and categories, only the highest level of function receives a 1; in others, two or more levels have scores of 1 because each describes competence that represents some minimal level of function.
  These screens are useful for indicating specifically how a person is performing at the present time. Therefore a higher score on the IADL would represent a higher functioning level. Highest score= 8 (high functioning), lowest score =0 (low functioning).
International physical activity questionnaire (IPARQ) | through study completion, an average of 1 year
  IPAQ assesses physical activity undertaken across a set of domains. The following values are used for the analysis: Walking = 3.3 METs, Moderate PA = 4.0 METs and Vigorous PA = 8.0 METs.
  Low= Individuals who not meet criteria for Categories 2 or 3 are considered to have a 'low' physical activity level.
  Moderate= a) 3 or more days of vigorous-intensity activity of at least 20 minutes per day b) 5 or more days of moderate-intensity activity and/or walking of at least 30 minutes per day c) 5 or more days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum Total physical activity of at least 600 MET-minutes/week. High= a) vigorous-intensity activity on at least 3 days achieving a minimum Total physical activity of at least 1500 MET-minutes/week b) 7 or more days of any combination of walking, moderate-intensity or vigorous-intensity activities achieving a minimum Total physical activity of at least 3000 MET-minutes/week.

CONTACTS AND LOCATIONS:
Overall Officials: Andy Pringle, PhD, Study Director — University of Derby
Locations (1):
- University of Derby, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barry BK, Carson RG. The consequences of resistance training for movement control in older adults. J Gerontol A Biol Sci Med Sci. 2004 Jul;59(7):730-54. doi: 10.1093/gerona/59.7.m730. PMID 15304540
- [Background] Carroll TJ, Barry B, Riek S, Carson RG. Resistance training enhances the stability of sensorimotor coordination. Proc Biol Sci. 2001 Feb 7;268(1464):221-7. doi: 10.1098/rspb.2000.1356. PMID 11217890
- [Background] Colado JC, Garcia-Masso X, Pellicer M, Alakhdar Y, Benavent J, Cabeza-Ruiz R. A comparison of elastic tubing and isotonic resistance exercises. Int J Sports Med. 2010 Nov;31(11):810-7. doi: 10.1055/s-0030-1262808. Epub 2010 Aug 11. PMID 20703977
- [Background] Colado JC, Triplett NT. Effects of a short-term resistance program using elastic bands versus weight machines for sedentary middle-aged women. J Strength Cond Res. 2008 Sep;22(5):1441-8. doi: 10.1519/JSC.0b013e31817ae67a. PMID 18714245
- [Background] Gardner MM, Buchner DM, Robertson MC, Campbell AJ. Practical implementation of an exercise-based falls prevention programme. Age Ageing. 2001 Jan;30(1):77-83. doi: 10.1093/ageing/30.1.77. PMID 11322678
- [Background] Gerards MHG, McCrum C, Mansfield A, Meijer K. Perturbation-based balance training for falls reduction among older adults: Current evidence and implications for clinical practice. Geriatr Gerontol Int. 2017 Dec;17(12):2294-2303. doi: 10.1111/ggi.13082. Epub 2017 Jun 16. PMID 28621015
- [Background] Lima FF, Camillo CA, Gobbo LA, Trevisan IB, Nascimento WBBM, Silva BSA, Lima MCS, Ramos D, Ramos EMC. Resistance Training using Low Cost Elastic Tubing is Equally Effective to Conventional Weight Machines in Middle-Aged to Older Healthy Adults: A Quasi-Randomized Controlled Clinical Trial. J Sports Sci Med. 2018 Mar 1;17(1):153-160. eCollection 2018 Mar. PMID 29535589
- [Background] Mansfield A, Aqui A, Centen A, Danells CJ, DePaul VG, Knorr S, Schinkel-Ivy A, Brooks D, Inness EL, McIlroy WE, Mochizuki G. Perturbation training to promote safe independent mobility post-stroke: study protocol for a randomized controlled trial. BMC Neurol. 2015 Jun 6;15:87. doi: 10.1186/s12883-015-0347-8. PMID 26048054
- [Background] Mansfield A, Peters AL, Liu BA, Maki BE. A perturbation-based balance training program for older adults: study protocol for a randomised controlled trial. BMC Geriatr. 2007 May 31;7:12. doi: 10.1186/1471-2318-7-12. PMID 17540020
- [Background] Youdas JW, Adams KE, Bertucci JE, Brooks KJ, Nelson MM, Hollman JH. Muscle activation levels of the gluteus maximus and medius during standing hip-joint strengthening exercises using elastic-tubing resistance. J Sport Rehabil. 2014 Feb;23(1):1-11. doi: 10.1123/jsr.2012-0082. Epub 2013 Aug 6. PMID 23921445
- See also: Department of Health- Physical activity guidelines — https://www.gov.uk/government/publications/physical-activity-guidelines-uk-chief-medical-officers-report
- See also: NHS Overview on Falls — https://www.nhs.uk/conditions/Falls/